CLINICAL TRIAL: NCT05278559
Title: Can Undetectable (Viral Load) = Untransmissible (Virus) Change the Life Course of Adolescents Living the HIV in Africa
Brief Title: Can Undetectable (Viral Load) = Untransmissible (Virus) Change the Life Course of Adolescents Living in Africa
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Centre for Sexual Health and HIV/AIDS Research Zimbabwe (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Other Study IDs: CeSHHAR
Record Dates: First submitted 2022-03-04; First posted 2022-03-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: HIV/AIDS
Keywords: AIDS - Acquired Immuno Dificiency Syndrome; ALHIV - Adolescents Living with HIV; CATS - Community Adolescents Treatment Supporters; DBS - Dried blood spot; MoHCC - Ministry of Health and Child Care; U=U - Undetectable = Untransimmisible; VL - Viral load
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescents living with HIV: - ALHIV with a viral load result of less than <1000 copies/mL and aged between 13-19 years

SUMMARY:
The scientific breakthrough related to Undetectable (viral load) = Untransmissible (virus) has had a major impact on motivation to take up and adhere to antiretroviral therapy among people living with HIV all over the world. The aim of the study is to work with MoHCC and other stakeholders to explore whether routine VL testing using DBS can provide sufficiently robust evidence of 'undetectability' to support introduction of U=U messaging in ALHIV. The study will provide scientific evidence on whether routine VL testing using DBS as available in LIC can provide sufficiently robust evidence of 'undetectability' and on the variability of an individual's virological response over 12 months. It will provide contextually orientated evidence to inform U=U messaging which has the potential to change the motivation of ALHIV to engage with their treatment and care.It will also explore responsible ways to disseminate this message to ALHIV living in Zimbabwe, and across the Southern African region.

DETAILED DESCRIPTION:
Rationale: Adolescents living with HIV (ALHIV) have the worst outcomes of all ages because of sub-optimal adherence driven by structural factors associated with poverty. This is exacerbated for adolescents by the limited opportunities to address mental health problems arising from the intersection of growing up in poverty and with HIV. The scientific breakthrough related to Undetectable (viral load) = Untransmissible (virus) has had a major impact on motivation to take up and adhere to antiretroviral therapy among people living with HIV all over the world. However, the discussion remains remarkably silent in high burden, low-income countries (LIC). Very few ALHIV in LIC are aware that having an undetectable viral load (VL) substantially reduces the risk of transmitting HIV to their sexual partners and children.

The aim of the study is to work with MoHCC and other stakeholders to explore whether routine VL testing using DBS can provide sufficiently robust evidence of 'undetectability' to support introduction of U=U messaging in ALHIV.

The specific objectives are:

1. To determine viral load fluctuation between routine annual VL testing and the extent to which annual VL using DBS reflects short term fluctuations that occur in the interim.
2. To determine what proportion of ALHIV with VL <1000 copies/uL on DBS have a plasma VL less than 200 copies/uL
3. To explore the reasons for and adolescent's understandings of fluctuations in VL and what a VL<1000 copies/mL means to ALHIV

Methods: This mixed method study will be conducted in conjunction with key stakeholders. We will enrol 300 ALHIV with a recent VL<1000 copies/uL in three HIV clinics in Harare and follow them for 12 months. Of these, 100 will be randomly selected to undergo repeat VL testing, using both DBS and plasma samples at enrolment, 6 and 12 months. A purposive sample of twenty will be selected for a longitudinal qualitative study. Additionally, up to eight participatory workshops will be conducted with key stakeholders over the course of the study to co-develop a 'safe' way to message U=U for LIC.

Potential impact: The study will provide scientific evidence on whether routine VL testing using DBS as available in LIC can provide sufficiently robust evidence of 'undetectability' and on the variability of an individual's virological response over 12 months. It will provide contextually orientated evidence to inform U=U messaging which has the potential to change the motivation of ALHIV to engage with their treatment and care.

ELIGIBILITY:
Inclusion Criteria:

* ALHIV aged 13-19 years who are aware of their HIV status for at least six months before enrolment (i.e., know the infection by its name and understand some of its implications).
* ART initiation of not less than 6 months.
* ALHIV accessing ART within the participating clinics.
* Healthcare workers with direct contact with ALHIV and have been involved in viral load result counselling in participating clinics.

Exclusion Criteria:

* Unable to provide informed assent/ and parental informed consent.
* Requires urgent medical attention or has severe mental health problems that would invalidate the informed assent/consent process or else contraindicate participation.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: We are recruiting adolescents aged 13-19 years both males and females. We are taking all the ALHIV in the age range even those who are married and have children.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
The study will provide scientific evidence on whether routine VL testing using DBS as available in LIC can provide sufficiently robust evidence of 'undetectability' and on the variability of an individual's virological response over 12 months. | One Year
  The study will explore the sensitivity of viral load testing so that decisions can be made on the best use of resources in optimizing the care and support that can be given to ALHIV in the region.
The study will assist in developing an evidence-base to support the U=U integration into standard of care. | Two years
  To unpack some of the key challenges that undermine ALHIV's engagement and there will be workshops with policy makers to discuss the findings and explore their perceptions on the feasibility of implementing policies related to U=U in this age group. Their views will be elicited around whether they consider there is 'safe' U=U messaging for LIC that could be implemented logistically, clinically and socially.

SECONDARY OUTCOMES:
It will generate peer-reviewed publications and educational resources. | Two years
  Working with the Ministry of Health and Child Care to develop locally appropriate ways of incorporating U=U into routine HIV treatment and care among ALHIV in Zimbabwe. We have already set up a technical working group comprising members from the MoHCC, AFRICAID ZVANDIRI and UNICEF. This was made possible through a UNICEF supported small-scale resource development project which is supporting development of resources for ALHIV to improve their HIV literacy and particularly their literacy related to viral load testing, which has been relatively recently introduced into routine HIV care in Zimbabwe.

CONTACTS AND LOCATIONS:
Overall Officials: Frances. M Cowan, Proffesor, Study Director — CeSHHAR Zimbabwe; Sarah Bernays, PhD, Study Chair — University of Sydney; Zivai Mupambireyi Nenguke, Principal Investigator — Centre for Sexual Health and HIV/AIDS Research Zimbabwe
Locations (1):
- Beatrice Road Infectious Hospital, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
We are going to be sharing Clinical results and overall study findings
Supporting Information: SAP, ICF, CSR, Analytic Code
Time Frame: As from January 2024
Access Criteria: Request access from Zivai

REFERENCES:
- [Background] Kouamou V, Manasa J, Katzenstein D, McGregor AM, Ndhlovu CE, Makadzange AT. Drug resistance and optimizing dolutegravir regimens for adolescents and young adults failing antiretroviral therapy. AIDS. 2019 Sep 1;33(11):1729-1737. doi: 10.1097/QAD.0000000000002284. PMID 31361272
- [Background] Casale M, Carlqvist A, Cluver L. Recent Interventions to Improve Retention in HIV Care and Adherence to Antiretroviral Treatment Among Adolescents and Youth: A Systematic Review. AIDS Patient Care STDS. 2019 Jun;33(6):237-252. doi: 10.1089/apc.2018.0320. PMID 31166783
- [Background] Martelli G, Antonucci R, Mukurasi A, Zepherine H, Nostlinger C. Adherence to antiretroviral treatment among children and adolescents in Tanzania: Comparison between pill count and viral load outcomes in a rural context of Mwanza region. PLoS One. 2019 Mar 21;14(3):e0214014. doi: 10.1371/journal.pone.0214014. eCollection 2019. PMID 30897131
- [Background] Boerma RS, Boender TS, Bussink AP, Calis JC, Bertagnolio S, Rinke de Wit TF, Boele van Hensbroek M, Sigaloff KC. Suboptimal Viral Suppression Rates Among HIV-Infected Children in Low- and Middle-Income Countries: A Meta-analysis. Clin Infect Dis. 2016 Dec 15;63(12):1645-1654. doi: 10.1093/cid/ciw645. Epub 2016 Sep 22. PMID 27660236
- [Background] Webb D, Cluver L, Luo C. Evolution or extinction? Paediatric and adolescent HIV responses in the Agenda 2030 era. J Int AIDS Soc. 2018 Feb;21 Suppl 1(Suppl Suppl 1):e25071. doi: 10.1002/jia2.25071. No abstract available. PMID 29485744
- [Background] Nachega JB, Sam-Agudu NA, Mofenson LM, Schechter M, Mellors JW. Achieving Viral Suppression in 90% of People Living With Human Immunodeficiency Virus on Antiretroviral Therapy in Low- and Middle-Income Countries: Progress, Challenges, and Opportunities. Clin Infect Dis. 2018 May 2;66(10):1487-1491. doi: 10.1093/cid/ciy008. PMID 29324994
- [Background] Mbirimtengerenji ND. Is HIV/AIDS epidemic outcome of poverty in sub-saharan Africa? Croat Med J. 2007 Oct;48(5):605-17. PMID 17948947
- [Background] Mavhu W, Willis N, Mufuka J, Bernays S, Tshuma M, Mangenah C, Maheswaran H, Mangezi W, Apollo T, Araya R, Weiss HA, Cowan FM. Effect of a differentiated service delivery model on virological failure in adolescents with HIV in Zimbabwe (Zvandiri): a cluster-randomised controlled trial. Lancet Glob Health. 2020 Feb;8(2):e264-e275. doi: 10.1016/S2214-109X(19)30526-1. Epub 2020 Jan 7. PMID 31924539
- [Background] Brown K, Williams DB, Kinchen S, Saito S, Radin E, Patel H, Low A, Delgado S, Mugurungi O, Musuka G, Tippett Barr BA, Nwankwo-Igomu EA, Ruangtragool L, Hakim AJ, Kalua T, Nyirenda R, Chipungu G, Auld A, Kim E, Payne D, Wadonda-Kabondo N, West C, Brennan E, Deutsch B, Worku A, Jonnalagadda S, Mulenga LB, Dzekedzeke K, Barradas DT, Cai H, Gupta S, Kamocha S, Riggs MA, Sachathep K, Kirungi W, Musinguzi J, Opio A, Biraro S, Bancroft E, Galbraith J, Kiyingi H, Farahani M, Hladik W, Nyangoma E, Ginindza C, Masangane Z, Mhlanga F, Mnisi Z, Munyaradzi P, Zwane A, Burke S, Kayigamba FB, Nuwagaba-Biribonwoha H, Sahabo R, Ao TT, Draghi C, Ryan C, Philip NM, Mosha F, Mulokozi A, Ntigiti P, Ramadhani AA, Somi GR, Makafu C, Mugisha V, Zelothe J, Lavilla K, Lowrance DW, Mdodo R, Gummerson E, Stupp P, Thin K, Frederix K, Davia S, Schwitters AM, McCracken SD, Duong YT, Hoos D, Parekh B, Justman JE, Voetsch AC. Status of HIV Epidemic Control Among Adolescent Girls and Young Women Aged 15-24 Years - Seven African Countries, 2015-2017. MMWR Morb Mortal Wkly Rep. 2018 Jan 12;67(1):29-32. doi: 10.15585/mmwr.mm6701a6. PMID 29329280
- [Background] Natukunda J, Kirabira P, Ong KIC, Shibanuma A, Jimba M. Virologic failure in HIV-positive adolescents with perfect adherence in Uganda: a cross-sectional study. Trop Med Health. 2019 Jan 17;47:8. doi: 10.1186/s41182-019-0135-z. eCollection 2019. PMID 30679930
- [Background] Ngarina M, Popenoe R, Kilewo C, Biberfeld G, Ekstrom AM. Reasons for poor adherence to antiretroviral therapy postnatally in HIV-1 infected women treated for their own health: experiences from the Mitra Plus study in Tanzania. BMC Public Health. 2013 May 7;13:450. doi: 10.1186/1471-2458-13-450. PMID 23647555
- [Background] The Lancet Hiv. U=U taking off in 2017. Lancet HIV. 2017 Nov;4(11):e475. doi: 10.1016/S2352-3018(17)30183-2. No abstract available. PMID 29096785
- [Background] Calabrese SK, Mayer KH. Providers should discuss U=U with all patients living with HIV. Lancet HIV. 2019 Apr;6(4):e211-e213. doi: 10.1016/S2352-3018(19)30030-X. Epub 2019 Feb 13. No abstract available. PMID 30772420
- [Background] Eisinger RW, Dieffenbach CW, Fauci AS. HIV Viral Load and Transmissibility of HIV Infection: Undetectable Equals Untransmittable. JAMA. 2019 Feb 5;321(5):451-452. doi: 10.1001/jama.2018.21167. No abstract available. PMID 30629090
- [Background] WHO. Dolutegravir (DTG) and the fixed dose combination of tenofovir/lamivudine/dolutegravir (TLD). Briefing Note, April 2018. Briefing Note [Internet]. 2018.
- [Background] Paul N, Ugwu R. Dolutegravir (DTG) Based Fixed Dose Combination (FDC) of Tenofovir/Lamivudine/Dolutegravir (TLD) and Viral Load Suppression in Children in Port Harcourt, Nigeria. Journal of Scientific Research and Reports. 2020:52-9.
- [Background] Ndashimye E, Arts EJ. The urgent need for more potent antiretroviral therapy in low-income countries to achieve UNAIDS 90-90-90 and complete eradication of AIDS by 2030. Infect Dis Poverty. 2019 Aug 2;8(1):63. doi: 10.1186/s40249-019-0573-1. PMID 31370888
- [Background] Sithole Z, Mbizvo E, Chonzi P, Mungati M, Juru TP, Shambira G, Gombe NT, Tshimanga M. Virological failure among adolescents on ART, Harare City, 2017- a case-control study. BMC Infect Dis. 2018 Sep 18;18(1):469. doi: 10.1186/s12879-018-3372-6. PMID 30227831
- [Background] Nyagadza B, Kudya N, Mbofana E, Masaka S, Garone D, Chen CY, Mulingwa A, Uzande C, Isaakidis P, Ndlovu Z. Scaling up HIV viral load monitoring in Manicaland, Zimbabwe: challenges and opportunities from the field. Public Health Action. 2019 Dec 21;9(4):177-181. doi: 10.5588/pha.19.0024. PMID 32042612
- [Background] Kilmarx PH, Simbi R. Progress and Challenges in Scaling Up Laboratory Monitoring of HIV Treatment. PLoS Med. 2016 Aug 23;13(8):e1002089. doi: 10.1371/journal.pmed.1002089. eCollection 2016 Aug. PMID 27551962
- [Background] Vreeman RC, McCoy BM, Lee S. Mental health challenges among adolescents living with HIV. J Int AIDS Soc. 2017 May 16;20(Suppl 3):21497. doi: 10.7448/IAS.20.4.21497. PMID 28530045
- [Background] Calabrese SK, Mayer KH. Stigma impedes HIV prevention by stifling patient-provider communication about U = U. J Int AIDS Soc. 2020 Jul;23(7):e25559. doi: 10.1002/jia2.25559. No abstract available. PMID 32686324
- [Background] Braun V, Clarke V. Using thematic analysis in psychology Qualitative Research in Psychology. 2006;3(2):77-101.
- [Background] Cohen MS, Chen YQ, McCauley M, Gamble T, Hosseinipour MC, Kumarasamy N, Hakim JG, Kumwenda J, Grinsztejn B, Pilotto JH, Godbole SV, Chariyalertsak S, Santos BR, Mayer KH, Hoffman IF, Eshleman SH, Piwowar-Manning E, Cottle L, Zhang XC, Makhema J, Mills LA, Panchia R, Faesen S, Eron J, Gallant J, Havlir D, Swindells S, Elharrar V, Burns D, Taha TE, Nielsen-Saines K, Celentano DD, Essex M, Hudelson SE, Redd AD, Fleming TR; HPTN 052 Study Team. Antiretroviral Therapy for the Prevention of HIV-1 Transmission. N Engl J Med. 2016 Sep 1;375(9):830-9. doi: 10.1056/NEJMoa1600693. Epub 2016 Jul 18. PMID 27424812
- [Background] Rodger AJ, Cambiano V, Bruun T, Vernazza P, Collins S, Degen O, Corbelli GM, Estrada V, Geretti AM, Beloukas A, Raben D, Coll P, Antinori A, Nwokolo N, Rieger A, Prins JM, Blaxhult A, Weber R, Van Eeden A, Brockmeyer NH, Clarke A, Del Romero Guerrero J, Raffi F, Bogner JR, Wandeler G, Gerstoft J, Gutierrez F, Brinkman K, Kitchen M, Ostergaard L, Leon A, Ristola M, Jessen H, Stellbrink HJ, Phillips AN, Lundgren J; PARTNER Study Group. Risk of HIV transmission through condomless sex in serodifferent gay couples with the HIV-positive partner taking suppressive antiretroviral therapy (PARTNER): final results of a multicentre, prospective, observational study. Lancet. 2019 Jun 15;393(10189):2428-2438. doi: 10.1016/S0140-6736(19)30418-0. Epub 2019 May 2. PMID 31056293
- [Background] Rodger AJ, Cambiano V, Bruun T, Vernazza P, Collins S, van Lunzen J, Corbelli GM, Estrada V, Geretti AM, Beloukas A, Asboe D, Viciana P, Gutierrez F, Clotet B, Pradier C, Gerstoft J, Weber R, Westling K, Wandeler G, Prins JM, Rieger A, Stoeckle M, Kummerle T, Bini T, Ammassari A, Gilson R, Krznaric I, Ristola M, Zangerle R, Handberg P, Antela A, Allan S, Phillips AN, Lundgren J; PARTNER Study Group. Sexual Activity Without Condoms and Risk of HIV Transmission in Serodifferent Couples When the HIV-Positive Partner Is Using Suppressive Antiretroviral Therapy. JAMA. 2016 Jul 12;316(2):171-81. doi: 10.1001/jama.2016.5148. PMID 27404185
- [Background] Bavinton BR, Pinto AN, Phanuphak N, Grinsztejn B, Prestage GP, Zablotska-Manos IB, Jin F, Fairley CK, Moore R, Roth N, Bloch M, Pell C, McNulty AM, Baker D, Hoy J, Tee BK, Templeton DJ, Cooper DA, Emery S, Kelleher A, Grulich AE; Opposites Attract Study Group. Viral suppression and HIV transmission in serodiscordant male couples: an international, prospective, observational, cohort study. Lancet HIV. 2018 Aug;5(8):e438-e447. doi: 10.1016/S2352-3018(18)30132-2. Epub 2018 Jul 17. PMID 30025681
- [Background] Chandra-Mouli V, Armstrong A, Amin A, Ferguson J. A pressing need to respond to the needs and sexual and reproductive health problems of adolescent girls living with HIV in low- and middle-income countries. J Int AIDS Soc. 2015 Dec 1;18(Suppl 5):20297. doi: 10.7448/IAS.18.6.20297. eCollection 2015. PMID 26643463
- [Background] 29. Alliance. IHA, Zvandiri. A. Supporting children, adolescents and young people living with HIV to start and stay on HIV treatment. Harare, Zimbabwe International HIV/AIDS Alliance; 2017.
- [Background] Willis N, Frewin L, Miller A, Dziwa C, Mavhu W, Cowan F. "My story"-HIV positive adolescents tell their story through film. Children and Youth Services Review. 2014;45:129-36

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/59/NCT05278559/Prot_SAP_000.pdf